CLINICAL TRIAL: NCT06441019
Title: Efficacy and Safety of HAIC in Combination With TQB2868 and Ramucirumab for Second-line Treatment of Advanced Hepatocellular Carcinoma: an Open, Single-arm Exploratory Study
Brief Title: Efficacy and Safety of HAIC in Combination With TQB2868 and Ramucirumab for Second-line Treatment of Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Chief physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2403292-19
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma，Bispecific Antibodies, HAIC, Ramucirumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC combined with TQB2868 and Ramucirumab (Experimental)
  Interventions: Drug: HAIC（Oxaliplatin+ Raltitrexed）、TQB2868、Ramucirumab

INTERVENTIONS:
Drug: HAIC（Oxaliplatin+ Raltitrexed）、TQB2868、Ramucirumab — The patient will receive combined treatment with HAIC, TQB2868, and Ramucirumab. After enrollment, the patient will undergo routine hepatic artery angiography via femoral artery catheterization and placement of a hepatic artery catheter，they will then receive 150ml of 5% sodium bicarbonate + Oxaliplatin (85mg/m2) for 4-6 hours + Raltitrexed (2mg/m2) for 2-4 hours . This will be done every 3-4 weeks for at least 2 cycles. Systemic treatment will be administered every 21 days, with TQB2868 injection given on the first day of each cycle (1-7 days after HAIC). The fixed dose of TQB2868 will be 300mg, and Ramucirumab will be given at a dose of 500mg (initial intravenous infusion for 60 minutes, followed by 30 minutes if tolerated).

SUMMARY:
In recent years, with the emergence of various new targeted and immunotherapy drugs, drug therapy for advanced Hepatocellular carcinoma has also seen continuous breakthroughs. The effective rate, progression free survival, and overall survival of advanced Hepatocellular carcinoma have all significantly improved. At present, internationally recognized first-line treatments available include atezolizumab+bevacizumab (T+A), lenvatinib, sorafenib, Durvalumab+tremelimumab, etc. However, the effective rate of first-line treatment has not exceeded 50%, and most patients face difficulties such as drug resistance or treatment failure. Second line treatment for Hepatocellular carcinoma still faces many difficulties and challenges. The aim of this study is to explore the effectiveness and safety of HAIC combined with TQB2868 and Ramucirumab in second-line treatment of advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female aged 18-80 years or older;
* Signed informed consent form;
* The investigator believes that the patient is capable of complying with the study protocol;
* Histologically or cytologically confirmed advanced hepatocellular carcinoma (HCC);
* Patients who have received first-line treatment for hepatocellular carcinoma and have treatment failure or intolerance;
* No prior treatment with HAIC including oxaliplatin;
* Prior treatment with tyrosine kinase inhibitors (TKIs) and/or immunotherapy is allowed;
* At least one measurable, untreated lesion according to RECIST 1.1 criteria;
* Availability of pretreatment tumor tissue sample, if available. If tumor tissue is not available (e.g., exhausted by previous diagnostic testing), the patient remains eligible for participation in the study;
* ECOG performance status of 0 or 1 within 14 days prior to enrollment;
* Child-Pugh class A or B ≤7 within 14 days prior to enrollment;
* Adequate hematologic and organ function;
* Any acute clinically significant treatment-related toxicity (from prior therapy) must have resolved to ≤Grade 1 prior to enrollment, except for alopecia;
* Negative HIV antibody test result at screening;
* Patients with active hepatitis B virus (HBV) infection: HBV DNA <2000 IU/mL obtained within 28 days prior to starting study treatment and at least 7 days of antiviral treatment (according to local standard of care, e.g., entecavir) prior to enrollment and willingness to continue treatment during the study; Patients with active hepatitis C virus (HCV) infection: HCV RNA <2000 IU/mL obtained within 28 days prior to starting study treatment and at least 7 days of antiviral treatment prior to enrollment and willingness to continue treatment during the study;
* Women of childbearing potential must have a negative pregnancy test (β-HCG) prior to initiation of treatment, and women of childbearing potential and men (who engage in sexual intercourse with women of childbearing potential) must agree to use effective contraception continuously during the treatment period and for 6 months after the last dose of treatment.

Exclusion Criteria:

* Previous treatment with HAIC containing oxaliplatin;
* Expected survival time less than 3 months
* History of meningitis;
* Current or past autoimmune diseases or immunodeficiency;
* Idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonia, or idiopathic pneumonia, or evidence of active pneumonia on screening computed tomography (CT) scan. Prior radiation pneumonitis in the radiation field (fibrosis) is allowed;
* Known active tuberculosis;
* Significant cardiovascular disease within 3 months prior to starting study treatment (e.g., New York Heart Association Class II or greater heart disease, myocardial infarction, or cerebrovascular accident), unstable arrhythmia, or unstable angina;
* History of congenital long QT syndrome or corrected QT interval >500ms (calculated using Fridericia's method) at screening;
* History of uncorrectable electrolyte disturbances such as serum potassium, calcium, or magnesium imbalances;
* Major surgery within 4 weeks prior to starting study treatment (excluding diagnostic procedures) or anticipation of need for major surgical procedure during the course of the study;
* History of malignancy other than HCC within 5 years prior to screening, unless the risk of recurrence or death from the previous malignancy is considered negligible (e.g., 5-year overall survival rate >90%) and adequately treated in situ cervical cancer, non-melanoma skin cancer, localized prostate cancer, in situ ductal carcinoma, or stage I uterine cancer;
* Severe infection within 4 weeks prior to starting study treatment, including but not limited to hospitalization for complications of infection, sepsis, or severe pneumonia;
* Treatment with therapeutic antibiotics orally or intravenously within 2 weeks prior to starting study treatment. Patients receiving prophylactic antibiotics (e.g., for prevention of urinary tract infection or exacerbation of chronic obstructive pulmonary disease) are eligible for participation in the study;
* Prior allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
* Receipt of attenuated live vaccines within 4 weeks prior to starting study treatment or anticipated need for such vaccines within 5 months after the last dose of PD-1 antibody therapy;
* Untreated or incompletely treated esophageal and/or gastric varices associated with bleeding or patients at high risk of bleeding;
* Concurrent HBV and HCV infection. Patients with a history of HCV infection but negative HCV RNA PCR results can be considered not infected with HCV;
* Symptomatic, untreated, or gradually progressing central nervous system (CNS) metastases;
* Inability to comply with follow-up or concurrent participation in another clinical trial that may interfere with this study;
* The investigator deems the patient unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 24 months
  The proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including complete response and partial response

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 2 years
  Time from enrollment to death
Disease Control Rate (DCR) | 6 months
  Disease Control Rate (DCR) based on RECIST v1.1 assessment
Progression-Free Survival (PFS) | Up to approximately 1 years
  Progression-Free Survival (PFS)
Incidence of Adverse Events and Treatment-Emergent Adverse Events | Up to approximately 2 years
  Safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China